CLINICAL TRIAL: NCT05929157
Title: A Crossover Bioavailability Clinical Trial of Parenteral Pyronaridine and Artesunate
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Ayola Akim ADEGNIKA, Professor, Centre de Recherche Médicale de Lambaréné
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: parP&A_22_1
Record Dates: First submitted 2023-06-16; First posted 2023-07-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Severe Malarial Treatment
MeSH Terms: interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: Phase I monocentric clinical trial with a two-armed crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artesunate-pyronaridine intravenous (Active Comparator)
  Interventions: Drug: artesunate-pyronaridine
- Artesunate-pyronaridine intramuscular (Active Comparator)
  Interventions: Drug: artesunate-pyronaridine

INTERVENTIONS:
Drug: artesunate-pyronaridine — Pyronaridine and Artesunate are antimalarial agents with a history of clinical use, and Artesunate has been used clinically in combination with other drugs also. The action of Artesunate is a rapid knock down of the parasites, after which, the drug is quickly cleared as it has a short systemic half-life. Pyronaridine is also rapidly effective in the short term but has a long blood half-life thus providing a more sustained schizonticidal effect.

SUMMARY:
The clinical trial is a Phase I monocentric clinical trial with a two-armed crossover design to evaluate the bioavailability of parenteral Pyronaridine and Artesunate.

Pyronaridine and Artesunate are antimalarial agents with a history of clinical use, and Artesunate has been used clinically in combination with other drugs also. The action of Artesunate is a rapid knock down of the parasites, after which, the drug is quickly cleared as it has a short systemic half-life. Pyronaridine is also rapidly effective in the short term but has a long blood half-life thus providing a more sustained schizonticidal effect.

12 study subjects will be included into the clinical trial after having signed the informed consent, being screened and judged to be eligible. 6 of them (group 1) will, on Day 0, be injected intravenously with 4 mg base/kg of Pyronaridine together with 4 mg/kg of Artesunate. The group 2 (the other 6 subjects) will on the same day (Day 0) be injected intramuscularly with the 4 mg base/kg of Pyronaridine together with 4 mg/kg of Artesunate (into separate sites) 8 weeks later group 1 will be injected intramuscularly with the same amount of Pyronaridine and Artesunate as on Day 0. Group 2 will also get the same amount as on Day 0 but this time the injection will be intravenously for group 2.

The primary objective is to assess the safety and tolerability by measuring (a) the proportion of subjects with adverse events (AEs) and serious adverse events (SAEs) throughout the study; (b) the proportion of subjects with solicited AEs 15 days after IMP injection; (c) the proportion of subjects with unsolicited AEs throughout the clinical trial. Further, the pharmacokinetics of both drugs will be determined.

DETAILED DESCRIPTION:
The clinical trial is a Phase I monocentric clinical trial with a two-armed crossover design to evaluate the bioavailability of parenteral Pyronaridine and Artesunate.

Pyronaridine and Artesunate are antimalarial agents with a history of clinical use, and Artesunate has been used clinically in combination with other drugs also. The action of Artesunate is a rapid knock down of the parasites, after which, the drug is quickly cleared as it has a short systemic half-life. Pyronaridine is also rapidly effective in the short term but has a long blood half-life thus providing a more sustained schizonticidal effect.

12 study subjects will be included into the clinical trial after having signed the informed consent, being screened and judged to be eligible. 6 of them (group 1) will, on Day 0, be injected intravenously with 4 mg base/kg of Pyronaridine together with 4 mg/kg of Artesunate. The group 2 (the other 6 subjects) will on the same day (Day 0) be injected intramuscularly with the 4 mg base/kg of Pyronaridine together with 4 mg/kg of Artesunate (into separate sites) 8 weeks later group 1 will be injected intramuscularly with the same amount of Pyronaridine and Artesunate as on Day 0. Group 2 will also get the same amount as on Day 0 but this time the injection will be intravenously for group 2.

The primary objective is to assess the safety and tolerability by measuring (a) the proportion of subjects with adverse events (AEs) and serious adverse events (SAEs) throughout the study; (b) the proportion of subjects with solicited AEs 15 days after IMP injection; (c) the proportion of subjects with unsolicited AEs throughout the clinical trial. Further, the pharmacokinetics of both drugs will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers aged 18-45 years with an asymptomatic Plasmodium falciparum infection.
* Able and willing (in the investigator's opinion) to comply with all trial requirements.
* General good health based on medical history and clinical examination.
* Written informed consent.
* Available to participate in follow-up for the duration of the trial (4 months in total).
* Reachable by phone during the whole trial period.
* Women only: Must agree to practice continuous effective contraception for the duration of the trial.

Exclusion Criteria:

* Pregnancy, lactation, or intention to become pregnant during the trial.
* Known HIV-, HBV- and HCV-infection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of injectable artesunate-pyronaridine | within the two week post injection
  To assess the safety and tolerability by measuring (a) the proportion of subjects with adverse events (AEs) and serious adverse events (SAEs) throughout the study; (b) the proportion of subjects with solicited AEs 15 days after IMP injection; (c) the proportion of subjects with unsolicited AEs throughout the clinical trial
Plasma level of Pyronaridine | iwithin the two week post injection
  Change in concentration of post IV/IM injection whole blood and plasma level of Pyronaridine will be summarized over time
Plasma level of Artesunate/dihydroartemisinin | within the two week post injection
  Change in concentration of post IV/IM injection plasma level of Artesunate/dihydroartemisinin will be summarized over time

SECONDARY OUTCOMES:
Pyronaridine area under the curve | within the two week post injection
  Pyronaridine area under the whole blood and plasma concentration versus time curves (AUC), over a 24-hour period, following dosing
Artesunate/dihydroartemisinin area under the curve | within the two week post injection
  Artesunate/dihydroartemisinin area under the plasma concentration versus time curve (AUC) , over a 24-hour period, following dosing

OTHER OUTCOMES:
Pyronaridine distribution | within the two week post injection
  Distribution of pyronaridine between red cells and plasma (calculated from whole blood and plasma concentration measurements) will be interesting to look at during and after infection (after the crossover point)
Pyronaridine metabolites | within the two week post injection
  If possible, Pyronaridine metabolites will be measured in the PK analysis, apart from the parent compound

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherches Médicales de Lammbaréné, Lambaréné, Moyen-Ogooué Province, Gabon

IPD SHARING:
Plan to Share IPD: No